CLINICAL TRIAL: NCT03317899
Title: A Randomized Controlled Trial Evaluating the Use of G-CSF After Plerixafor-Mobilized Autologous Stem Cell Transplant (Auto HSCT)
Brief Title: Stem Cell Transplant With or Without Tbo-filgrastim in Treating Patients With Multiple Myeloma or Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17D.404; JT 10928 (Other: JeffTrial Number)
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Non-Hodgkin's Lymphoma; Plasma Cell Myeloma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — Stem Cell Transplantation; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group I (auto HSCT tbo-filgrastim) (Experimental): Beginning on day 3 after auto Hematopoietic Cell Transplantation (HSCT), patients receive tbo-filgrastim SC daily for 12-14 days.
  Interventions: Procedure: Hematopoietic Cell Transplantation; Drug: Tbo-filgrastim; Other: Laboratory Biomarker Analysis
- Group II (auto HSCT) (Experimental): Patients undergo auto Hematopoietic Cell Transplantation (HSCT).
  Interventions: Procedure: Hematopoietic Cell Transplantation; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Hematopoietic Cell Transplantation — Undergo auto HSCT
Drug: Tbo-filgrastim — Given subcutaneously
  Other Names: Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Granix
  Arms: Group I (auto HSCT tbo-filgrastim)
Other: Laboratory Biomarker Analysis — Correlative Studies

SUMMARY:
This phase II trial studies how well stem cell transplant with or without tbo-filgrastim works in treating patients with multiple myeloma or non-Hodgkin lymphoma. Eliminating the use of tbo-filgrastim after transplant may still help maintain a similar time to discharge.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate non-inferiority in the number of days to discharge readiness after a granulocyte colony-stimulating factor (G-CSF) + plerixafor-mobilized autologous stem cell transplant in patients receiving versus not receiving post-transplant growth factor support.

SECONDARY OBJECTIVE:

I. To compare days to absolute neutrophil count (ANC) > 500, days to platelet engraftment, febrile days, days of febrile neutropenia, documented infections, and number of antibiotic days in patients receiving versus not receiving post-transplant growth factor support.

EXPLORATORY OBJECTIVE:

I. To evaluate immunological recovery (lymphocyte number including CD 3/4 and CD3/8 T cell subsets) at day + 60 in patients receiving versus not receiving post-transplant growth factor support.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing autologous stem cell transplant for one of the following diagnoses:

  * Multiple myeloma
  * Non-Hodgkin lymphoma
* Karnofsky performance status of >= 70%
* Patients must meet the Thomas Jefferson University Hospital (TJUH) bone marrow transplant (BMT) standard of procedure (SOP) guidelines for "Patient Criteria for Autologous HSCT"
* Left ventricular ejection fraction (LVEF) of ≥ 40%
* Adjusted Carbon monoxide diffusing capability (DLCO) > 45% of predicted corrected for hemoglobin
* Serum bilirubin < 1.8
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2.5 X upper limit of normal
* Serum creatinine =< 2.0 mg/dl and/or creatinine clearance of > 40 ml/min (excludes multiple myeloma patients receiving high dose melphalan conditioning)
* Willingness to use contraception if childbearing potential
* Has the ability to give informed consent, or for cognitively or decisionally impaired individuals (vulnerable population), the availability of a family member or guardian to give consent and assist in the consent process
* Life expectancy of > 12 months (exclusive of the disease for which the auto HSCT is being performed)
* Patients must have undergone stem cell mobilization with the combination of G-CSF and plerixafor as per TJUH BMT SOP guidelines
* Collection of an adequate number of CD34+ stem cells, i.e. >= 4-6 x 10^6/kg from apheresis

Exclusion Criteria:

* Uncontrolled human immunodeficiency virus (HIV)
* Uncontrolled bacterial infection
* Active central nervous system (CNS) disease
* Pregnancy or lactation
* Evidence of another malignancy, exclusive of a skin cancer that requires only local treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Grosso, DNP, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group I (auto HSCT tbo-filgrastim) | Group II (auto HSCT)
Started | 38 | 39
Completed | 32 | 30
Not Completed | 6 | 9
Not completed — Death | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Auto HSCT Tbo-filgrastim) | Group II (Auto HSCT) | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 20 | 49
  >=65 years | 9 | 19 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 20 | 32
  Male | 26 | 19 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 33 | 37 | 70
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 24 | 27 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Days to Discharge
Description: Will compare days to discharge readiness between the two groups.
Time Frame: Up to 60 days
Measure: Median (Full Range); unit: days
Arm/Group | Group I (auto HSCT tbo-filgrastim) | Group II (auto HSCT)
Number analyzed (Participants) | 38 | 39
days | 11 [8 to 26] | 15 [11 to 29]
Statistical Analysis 1: Comparison: Group I (auto HSCT tbo-filgrastim) vs Group II (auto HSCT); Test type: Non-Inferiority — Weibull accelerated failure time model; adjusted for disease type and stem cell collection days; non-inferiority declared if 90% CI upper bound for acceleration factor < 1.133 (≤13.3% increase in discharge readiness time); one-sided α = 0.05; sample size for ~80% power; O'Brien-Fleming futility boundary applied; p = 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Median Days Post Autologous Hematopoietic Cell Transplantation (Auto HSCT) to Neutrophil Engraftment
Description: Will be defined as absolute neutrophil count > 500 x 10^9/L x 3 days. Day of engraftment is the first of the 3 days of absolute neutrophil count > 500 x 10^9/L.
Time Frame: Up to 60 days
Measure: Median (Full Range); unit: days
Arm/Group | Group I (auto HSCT tbo-filgrastim) | Group II (auto HSCT)
Number analyzed (Participants) | 38 | 39
days | 11 [8 to 13] | 13 [11 to 16]
Statistical Analysis 1: Comparison: Group I (auto HSCT tbo-filgrastim) vs Group II (auto HSCT); Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Median Days Post Auto HSCT to Platelet Engraftment
Description: Will be defined as date platelet greater than or equal to 20 x 10^9 /L without a platelet transfusion within the last 7 days.
Time Frame: Up to 60 days
Measure: Median (Full Range); unit: days
Arm/Group | Group I (auto HSCT tbo-filgrastim) | Group II (auto HSCT)
Number analyzed (Participants) | 38 | 39
days | 19 [16 to 25] | 19 [16 to 27]
Statistical Analysis 1: Comparison: Group I (auto HSCT tbo-filgrastim) vs Group II (auto HSCT); Test type: Other; p = 0.578, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Percentage of Participants With Engraftment Syndrome
Description: Will be defined by the Maiolino Criteria. Will be summarized by treatment arm and compared using a chi-square test
Time Frame: Up to 60 days
Measure: Number; unit: percentage of participants
Arm/Group | Group I (auto HSCT tbo-filgrastim) | Group II (auto HSCT)
Number analyzed (Participants) | 38 | 39
percentage of participants | 48.6 | 60
Statistical Analysis 1: Comparison: Group I (auto HSCT tbo-filgrastim) vs Group II (auto HSCT); Test type: Other; p = 0.337, Chi-squared

5. Secondary Outcome: Median Number of Febrile Days During the Auto HSCT Inpatient Stay
Description: Will be summarized by treatment arm and compared using Wilcoxon rank sum tests
Time Frame: Up to 60 days
Population: This data set was not reported. Upon further inspection into the subject data, there were few infections and most of the fevers were from neutropenia. No qualifying infections or fevers were reported to fit this specific criteria. Therefore, the numbers are presented as zero for both arms. Specific adverse event reporting data can be found in more detail in the AE/SAE section of this record.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (auto HSCT tbo-filgrastim) | Group II (auto HSCT)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Median Number of Days of Febrile Neutropenia During the Auto HSCT Inpatient Stay
Description: Will be summarized by treatment arm and compared using Wilcoxon rank sum tests.
Time Frame: Up to 60 days
Measure: Median (Full Range); unit: days of inpatient febrile neutropenia
Arm/Group | Group I (auto HSCT tbo-filgrastim) | Group II (auto HSCT)
Number analyzed (Participants) | 38 | 39
days of inpatient febrile neutropenia | 2 [0 to 6] | 4 [1 to 9]
Statistical Analysis 1: Comparison: Group I (auto HSCT tbo-filgrastim) vs Group II (auto HSCT); Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Median Number of Documented Infections Treatment During the Auto HSCT Inpatient Stay
Description: Will be defined as a positive blood culture not ultimately deemed to be due to a contaminant
Time Frame: Up to 60 days
Measure: Median (Full Range); unit: documented inpatient stay infections
Arm/Group | Group I (auto HSCT tbo-filgrastim) | Group II (auto HSCT)
Number analyzed (Participants) | 38 | 39
documented inpatient stay infections | 0 [0 to 3] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Group I (auto HSCT tbo-filgrastim) vs Group II (auto HSCT); Test type: Other; p = 0.936, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Median Number of Antibiotic Days During the Auto HSCT Inpatient Stay
Description: Will be summarized by treatment arm and compared using Wilcoxon rank sum tests.
Time Frame: Up to 60 days
Measure: Median (Full Range); unit: antibiotic inpatient days
Arm/Group | Group I (auto HSCT tbo-filgrastim) | Group II (auto HSCT)
Number analyzed (Participants) | 38 | 39
antibiotic inpatient days | 4 [0 to 14] | 7 [2 to 16]
Statistical Analysis 1: Comparison: Group I (auto HSCT tbo-filgrastim) vs Group II (auto HSCT); Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Percentage of Participants Receiving Corticosteroids
Description: will be presented as percentage of number of subjects who had the treatment
Time Frame: Up to 60 days
Population: Protocol initially stated that median number of days on corticosteroids will be summarized by treatment arm and compared using Wilcoxon rank sum tests up to 60 days; data reported as Steroids initiated percentage
Measure: Number; unit: percentage of patients
Arm/Group | Group I (auto HSCT tbo-filgrastim) | Group II (auto HSCT)
Number analyzed (Participants) | 38 | 39
percentage of patients | 31.4 | 51.4
Statistical Analysis 1: Comparison: Group I (auto HSCT tbo-filgrastim) vs Group II (auto HSCT); Test type: Other; p = 0.089, Chi-squared

10. Secondary Outcome: Percentage of Participants With Post Discharge Granulocyte Colony-stimulating Factor Administrations Through Day +60 Post Auto HSCT
Description: will be presented as percentage of number of subjects who had the treatment
Time Frame: Up to 60 days
Population: Protocol initially stated that number of post discharge granulocyte colony-stimulating factor administrations through day +60 post auto HSCT will be summarized by treatment arm and compared using Wilcoxon rank sum tests up to 60 days; data available is reported as reported as number with G-CSF
Measure: Number; unit: Percentage of Participants
Arm/Group | Group I (auto HSCT tbo-filgrastim) | Group II (auto HSCT)
Number analyzed (Participants) | 38 | 39
Percentage of Participants | 5.7 | 8.6
Statistical Analysis 1: Comparison: Group I (auto HSCT tbo-filgrastim) vs Group II (auto HSCT); Test type: Other; p = 0.645, Chi-squared

ADVERSE EVENTS:
Time Frame: Patients will be followed for adverse events for 60 days post-Auto HSCT
Arm/Group | Group I (auto HSCT tbo-filgrastim) | Group II (auto HSCT)
All-Cause Mortality (participants affected / at risk) | 6/37 | 9/39
Serious Adverse Events (participants affected / at risk) | 6/37 | 10/39
Other Adverse Events (participants affected / at risk) | 37/37 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (auto HSCT tbo-filgrastim) (N=37) | Group II (auto HSCT) (N=39)
Hypoxia (Vascular disorders) | 5 (5) | 1 (1)
Hypoglycemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Asparte aminotransferase (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
syncope (Vascular disorders) | 1 (1) | 0 (0)
Typhlitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
hypotension (Vascular disorders) | 1 (1) | 2 (2)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
infection/infestation (General disorders) | 0 (0) | 1 (1)
Engraftment syndrome (Immune system disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Urinary tract infection (Hepatobiliary disorders) | 0 (0) | 1 (1)
AST increase (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (auto HSCT tbo-filgrastim) (N=37) | Group II (auto HSCT) (N=39)
Atrial Fibrillation (grade1) (Cardiac disorders) | 2 (2) | 0 (0)
Atrial Fibrillation ( grade 2) (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Grade 3) (Cardiac disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Aortic Stenosis Grade 2 (Cardiac disorders) | 0 (0) | 1 (1)
asymptomatic LV dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
B12 deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1)
chest pain grade 1 (Cardiac disorders) | 2 (2) | 0 (0)
chest pain grade 2 (Cardiac disorders) | 2 (2) | 1 (1)
deep vein thrombosis grade 1 (Cardiac disorders) | 2 (2) | 2 (2)
deep vein thrombosis grade 2 (Cardiac disorders) | 2 (2) | 1 (1)
dyslipidemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
edema grade 1 (Cardiac disorders) | 20 (20) | 12 (12)
edema grade 2 (Cardiac disorders) | 0 (0) | 1 (1)
Hypercholesterolemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
hyperlipidemia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
hypergylcemia (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
hypertension grade 1 (Cardiac disorders) | 16 (26) | 13 (13)
hypertension grade 2 (Cardiac disorders) | 1 (1) | 0 (0)
hypotension Grade 1 (Cardiac disorders) | 18 (18) | 7 (7)
hypotension grade 2 (Cardiac disorders) | 3 (3) | 2 (2)
hypotension grade 3 (Cardiac disorders) | 1 (1) | 2 (2)
hypotension grade 4 (Cardiac disorders) | 0 (0) | 1 (1)
hypoxia grade 2 (Cardiac disorders) | 1 (1) | 1 (1)
hypoxia grade 3 (Cardiac disorders) | 5 (5) | 1 (1)
hypoxia grade 5 (Cardiac disorders) | 0 (0) | 1 (1)
Infusion Related Reaction Grade 1 (Cardiac disorders) | 1 (1) | 2 (2)
tacycardia (Cardiac disorders) | 15 (15) | 15 (15)
infusion related reaction grade 2 (Cardiac disorders) | 1 (1) | 1 (1)
murmur (Cardiac disorders) | 3 (3) | 3 (3)
normocytic anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
palpitations (Cardiac disorders) | 3 (3) | 3 (3)
supraventriculartachycardia grade2 (Cardiac disorders) | 1 (1) | 0 (0)
supraventriculartachycardia grade 4 (Cardiac disorders) | 1 (1) | 0 (0)
stroke grade 4 (Cardiac disorders) | 0 (0) | 1 (1)
PERICATHETER THROMBUS (Surgical and medical procedures) | 2 (2) | 0 (0)
premature ventricular contractions (Cardiac disorders) | 0 (0) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
thromboembolic event grade1 (Cardiac disorders) | 3 (3) | 0 (0)
thromboembolic event grade 2 (Cardiac disorders) | 1 (1) | 1 (1)
thromboembolic event grade 4 (Cardiac disorders) | 0 (0) | 1 (1)
abdominal cramps (Gastrointestinal disorders) | 1 (1) | 1 (1)
abdominal pain grade 1 (Gastrointestinal disorders) | 17 (17) | 13 (13)
abdominal pain grade 2 (General disorders) | 1 (1) | 2 (2)
abdominal swelling (Gastrointestinal disorders) | 3 (3) | 2 (2)
altered taste (Gastrointestinal disorders) | 1 (1) | 0 (0)
anorexia grade 2 (Gastrointestinal disorders) | 1 (1) | 0 (0)
belching (Gastrointestinal disorders) | 0 (0) | 2 (2)
blisters in mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
bloating (Gastrointestinal disorders) | 7 (7) | 2 (2)
bloody stools (Gastrointestinal disorders) | 0 (0) | 1 (1)
c-diff infection (Gastrointestinal disorders) | 0 (0) | 1 (1)
colitis grade 1 (Gastrointestinal disorders) | 2 (2) | 2 (2)
colitis grade 2 (Gastrointestinal disorders) | 1 (1) | 0 (0)
colon polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 15 (15) | 18 (18)
DIARRHEA Grade 1 (Gastrointestinal disorders) | 31 (31) | 21 (21)
DIARRHEA Grade 2 (Gastrointestinal disorders) | 1 (1) | 4 (4)
diverticulitis grade 1 (Gastrointestinal disorders) | 2 (2) | 0 (0)
diverticulitis grade 2 (General disorders) | 1 (1) | 0 (0)
dry mouth (Gastrointestinal disorders) | 5 (5) | 6 (6)
DYSGEUSIA (Gastrointestinal disorders) | 4 (4) | 0 (0)
elevated ALT grade 1 (Gastrointestinal disorders) | 1 (1) | 0 (0)
elevated ALT grade 2 (Gastrointestinal disorders) | 0 (0) | 1 (1)
dyspepsia grade 2 (Gastrointestinal disorders) | 0 (0) | 1 (1)
elevated LDH (Gastrointestinal disorders) | 1 (1) | 0 (0)
elevated liver function test grade 2 (Gastrointestinal disorders) | 1 (1) | 0 (0)
EPIGASTRIC BURNING (Gastrointestinal disorders) | 1 (1) | 0 (0)
EPIGASTRIC TIGHTNESS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ESOPHAGEAL SPASMS grade 2 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence grade 1 (Gastrointestinal disorders) | 7 (7) | 3 (3)
Flatulence grade 2 (Gastrointestinal disorders) | 0 (0) | 1 (1)
gas distention (Gastrointestinal disorders) | 6 (6) | 8 (8)
gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
GERD (Gastrointestinal disorders) | 12 (12) | 11 (11)
HEMORRHOIDS (Gastrointestinal disorders) | 2 (2) | 2 (2)
HEPTOBILIARY DISORDER Grade 3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
hiccups (Gastrointestinal disorders) | 4 (4) | 1 (1)
irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
ICTERUS/JAUNDICE (Gastrointestinal disorders) | 1 (1) | 0 (0)
indigestion (Gastrointestinal disorders) | 1 (1) | 2 (2)
JAW TENDERNESS (Gastrointestinal disorders) | 1 (1) | 0 (0)
LOWER GI HEMORRHAGE grade 3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
mouth sores (Gastrointestinal disorders) | 0 (0) | 1 (1)
MUCOSITIS Grade 1 (Gastrointestinal disorders) | 14 (14) | 14 (14)
MUCOSITIS Grade 2 (Gastrointestinal disorders) | 1 (1) | 3 (3)
MUCOSITIS Grade 3 (Gastrointestinal disorders) | 1 (1) | 1 (1)
nausea grade 1 (Gastrointestinal disorders) | 30 (30) | 32 (32)
nausea grade 2 (Gastrointestinal disorders) | 1 (1) | 0 (0)
obesity (Gastrointestinal disorders) | 3 (3) | 5 (5)
Ostomy prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
SMALL BOWEL OBSTRUCTION Grade 2 (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestine obstruction Grade 3 (Gastrointestinal disorders) | 1 (1) | 1 (1)
TROUBLE SWALLOWING (Gastrointestinal disorders) | 1 (1) | 0 (0)
TYPHILITIS Grade 3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
ULCER SUBLINGUAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
vomiting grade 1 (Gastrointestinal disorders) | 16 (16) | 13 (13)
vomiting grade 2 (Gastrointestinal disorders) | 1 (1) | 0 (0)
alopecia (Endocrine disorders) | 15 (15) | 8 (8)
DECREASED/ LOSS OF APPETITE grade 1 (Endocrine disorders) | 24 (24) | 17 (17)
DECREASED/ LOSS OF APPETITE grade 2 (Endocrine disorders) | 1 (1) | 1 (1)
DIABETES (Endocrine disorders) | 7 (7) | 2 (2)
HYPOGLYCEMIA (Endocrine disorders) | 2 (2) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 2 (2)
LYMPHEDEMA (Immune system disorders) | 2 (2) | 0 (0)
WEIGHT GAIN (Endocrine disorders) | 2 (2) | 1 (1)
alkaline grade 2 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
allergies (Immune system disorders) | 0 (0) | 2 (2)
chills grade 1 (Immune system disorders) | 10 (10) | 13 (13)
chills grade 2 (Immune system disorders) | 1 (1) | 0 (0)
fever grade 1 (Immune system disorders) | 27 (27) | 26 (26)
fever grade 2 (Immune system disorders) | 0 (0) | 2 (2)
HYPOGAMMAGLOBULINEMIA (Immune system disorders) | 1 (1) | 0 (0)
infection grade 1 (Infections and infestations) | 1 (1) | 0 (0)
infection grade 2 (Infections and infestations) | 2 (2) | 0 (0)
infection grade 3 (Infections and infestations) | 3 (3) | 1 (1)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
BURNING-TOES (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
DUPUYTRENS DISEASE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
EDEMATOUS SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
FOLLICULITIS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
IV SITE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PRURITIS-ITCH GRADE 1 (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7)
PRURITIS-ITCH GRADE 2 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Grade 1 (Skin and subcutaneous tissue disorders) | 17 (17) | 12 (12)
Rash Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
SUBCUTANEOUS TISSUE DISORDER (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
wound (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
enlarged lymph nodes (Immune system disorders) | 2 (2) | 0 (0)
weight loss (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
ARM PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ARM TWITCHING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12 (12) | 5 (5)
ARTHRITIS R HIP (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BACK PAIN Grade 1 (Musculoskeletal and connective tissue disorders) | 3 (3) | 12 (12)
BACK PAIN Grade 2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 10 (10)
BLIND IN LEFT EYE (Eye disorders) | 0 (0) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
BRUISES/BLEEDS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 1 (1)
CHEST TIGHTNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
CHIN NUMBNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
EYE DISCHARGE (Eye disorders) | 0 (0) | 1 (1)
COMPRESSION FRACTURE (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
FACIAL SWELLING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 1 (1)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 1 (1)
EXTREMITY WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
EYE IRRITATION (Eye disorders) | 0 (0) | 2 (2)
EYE SWELLING (Eye disorders) | 0 (0) | 2 (2)
Fall grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
FACIAL FLUSHING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
FACIAL ASYMMETRY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 32 (32) | 13 (13)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
GAIT PROBLEM Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
GAIT PROBLEM Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
HAND SPASM (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HEARING LOSS (Ear and labyrinth disorders) | 2 (2) | 3 (3)
HEEL SPUR PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HIP PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HYPOMAGNESEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
JAW PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
JOINT SWELLING Grade 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
JOINT SWELLING Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
KNEE PAIN Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
KYPHOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
L HAND SWELLING/TENDERNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LEFT EAR FULLNESS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
LEFT GAZE PALSY (Eye disorders) | 1 (1) | 0 (0)
LEG CRAMPS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
LEG WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
NECK STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN-PICC SITE (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
PELVIS-BURNING PRESSURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PERI-ANAL ITCHING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PETECHHIAE OF BILATERAL CALVES (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
RED EYE (Eye disorders) | 0 (0) | 1 (1)
R HAND SWELLING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
R THIGH PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RIB PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SORENESS BILATERAL LEGS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
STYE OF RIGHT EYELID (Eye disorders) | 0 (0) | 1 (1)
SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
WEAKNESS GRADE 1 (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7)
WEAKNESS GRADE 2 (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
ADHD (Nervous system disorders) | 1 (1) | 0 (0)
ANXIETY GRADE 1 (Nervous system disorders) | 8 (8) | 10 (10)
ANXIETY GRADE 2 (Nervous system disorders) | 1 (1) | 0 (0)
AGITATION GRADE 2 (Nervous system disorders) | 0 (0) | 1 (1)
BIPOLAR DSORDER (Nervous system disorders) | 1 (1) | 0 (0)
BLURRED VISION (Eye disorders) | 1 (1) | 0 (0)
CONJUNCTIVITIS (Eye disorders) | 1 (1) | 0 (0)
CONFUSION GRADE 1 (Nervous system disorders) | 0 (0) | 3 (3)
CONFUSION GRADE 2 (Nervous system disorders) | 0 (0) | 1 (1)
DEPRESSION (Nervous system disorders) | 4 (4) | 6 (6)
DIAPHORESIS (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS GRADE 1 (Nervous system disorders) | 9 (9) | 8 (8)
DIZZINESS GRADE 2 (Nervous system disorders) | 0 (0) | 1 (1)
DOUBLE VISION (Eye disorders) | 1 (1) | 1 (1)
DRY EYE (Eye disorders) | 1 (1) | 0 (0)
EYE DISCHARGE (Eye disorders) | 1 (1) | 0 (0)
FLAT AFFECT (Nervous system disorders) | 0 (0) | 1 (1)
FLUSHING (Nervous system disorders) | 0 (0) | 1 (1)
GLAUCOMA (Eye disorders) | 0 (0) | 1 (1)
HALLUCINATIONS GRADE 1 (Nervous system disorders) | 1 (1) | 0 (0)
HALLUCINATIONS GRADE 2 (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 9 (9) | 4 (4)
HERPETIC POLYNEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1)
HOT FLASHES (Endocrine disorders) | 0 (0) | 1 (1)
INSOMNIA (General disorders) | 14 (14) | 4 (4)
INSOMNIA GRADE 2 (General disorders) | 0 (0) | 1 (1)
LEFT FACIAL DROOP (General disorders) | 0 (0) | 1 (1)
LIGHTHEADED GRADE 1 (Nervous system disorders) | 2 (2) | 3 (3)
LIGHTHEADED GRADE 2 (Nervous system disorders) | 0 (0) | 1 (1)
LIP QUIVER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MAJOR DEPRESSIVE DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
MIGRAINE (Nervous system disorders) | 1 (1) | 0 (0)
NEUROPATHY GRADE 1 (Nervous system disorders) | 13 (13) | 8 (8)
NEUROPATHY GRADE 2 (Nervous system disorders) | 3 (3) | 1 (1)
NUMBNESS (Nervous system disorders) | 0 (0) | 1 (1)
NYSTAGMUS GRADE 2 (Nervous system disorders) | 0 (0) | 1 (1)
PALE CONJUNCTIVAE (Eye disorders) | 1 (1) | 0 (0)
PERIPHERAL NEUROPATHY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
PAIN/MYALGIA GRADE 1 (Nervous system disorders) | 12 (12) | 6 (6)
PAIN/MYALGIA GRADE 2 (Nervous system disorders) | 0 (0) | 3 (3)
PLOYNEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
PRESYNCOPE GRADE 2 (Nervous system disorders) | 1 (1) | 0 (0)
RIGHT FACIAL DROOP (General disorders) | 0 (0) | 1 (1)
RIGORS GRADE 1 (Nervous system disorders) | 1 (1) | 3 (3)
RIGORS GRADE 2 (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE GRADE 3 (Nervous system disorders) | 1 (1) | 0 (0)
SCIATIC PAIN (Nervous system disorders) | 0 (0) | 1 (1)
SLURRED SPEECH (Nervous system disorders) | 0 (0) | 1 (1)
TINNITUS (Nervous system disorders) | 0 (0) | 2 (2)
TREMORS (Nervous system disorders) | 1 (1) | 1 (1)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 (1) | 0 (0)
FIBROIDS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PENILE BLEEDING (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PENILE RASH (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PRURITIS-VAGINAL (Reproductive system and breast disorders) | 1 (1) | 1 (1)
VAGINAL SPOTTING/CRAMPS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
SCROTAL EDEMA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
BPH (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ATELECTASIS BILATERAL LOWER LOBE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 8 (8)
COURSE BREATH SOUNDS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CRACKLES @ BASES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DEEP BREATHING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNEA ON EXERTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
EXERCISE INDUCED ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Obstructive Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMONITIS GRADE 2 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
POST NASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
POST NASAL DRIP GRADE 2 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM GRADE 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RALES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RHINITIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
TACHYPNEA GRADE 1 (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
TACHYPNEA GRADE 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
BLADDER OUTLET OBSTRUCTION GRADE 2 (Renal and urinary disorders) | 1 (1) | 0 (0)
AKI (Renal and urinary disorders) | 0 (0) | 1 (1)
BPH (Renal and urinary disorders) | 12 (12) | 0 (0)
CKD (Renal and urinary disorders) | 1 (1) | 1 (1)
CKD GRADE 2 (Renal and urinary disorders) | 2 (2) | 0 (0)
DEHYDRATION (Renal and urinary disorders) | 2 (2) | 2 (2)
DIFFICULTY URINATING (Renal and urinary disorders) | 1 (1) | 0 (0)
DYSURIA GRADE 1 (Renal and urinary disorders) | 3 (3) | 3 (3)
DYSURIA GRADE 2 (Renal and urinary disorders) | 1 (1) | 0 (0)
HEMATURIA GRADE 1 (Renal and urinary disorders) | 1 (1) | 1 (1)
HEMATURIA GRADE 2 (Renal and urinary disorders) | 1 (1) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
HYPERKALEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HYPERVOLEMIA GRADE 2 (Renal and urinary disorders) | 1 (1) | 0 (0)
INCONTINENCE (Renal and urinary disorders) | 1 (1) | 1 (1)
HYPOKALEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
LUPUS NEPHRITIS (Renal and urinary disorders) | 1 (1) | 0 (0)
METABOLIC ACIDOSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1)
NOCTURIA (Renal and urinary disorders) | 13 (13) | 4 (4)
MYELOMA KIDNEY DISEASE (Renal and urinary disorders) | 1 (1) | 0 (0)
OVERACTIVE BLADDER (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL DISORDER (Renal and urinary disorders) | 2 (2) | 0 (0)
URINARY HESITANCY (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY FREQUENCY (Renal and urinary disorders) | 6 (6) | 5 (5)
URINARY RETENTION (Renal and urinary disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT03317899/Prot_SAP_000.pdf